CLINICAL TRIAL: NCT03500978
Title: Factors Predicting Ineffective Contraception Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HD091927; 1R21HD091927 (NIH)
Record Dates: First submitted 2018-04-02; First posted 2018-04-18 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Contraception Behavior
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Intervention Model Description: Two group (behavioral intervention vs. no treatment) randomized trial with a pre-intervention and 10- and 14-week post-intervention assessment phases.
Who Masked: Outcomes Assessor
Masking Description: Randomization occurs after the baseline assessment, so the assessor is blinded to study condition. Follow-up assessments of outcome are completed by study personnel who are blinded to intervention (i.e., they had no part in the intervention and no access to the randomization schedule). An electronic research management system (RedCAP) is used to deliver the random assignments to the interventionist digitally after baseline is completed. None of the data collection or intervention staff have access to the database underlying the random assignment in RedCAP. The randomization schedule was established by the biostatistician, who has no role in the data collection or intervention delivery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer CBT Intervention (Experimental): Women allocated to the peer-specialist delivered CBT intervention group will be mailed an intervention workbook (CBT exercises) and have their first telephone-based intervention session scheduled. The CBT intervention group will receive 8 telephone-based CBT intervention sessions (over 9 weeks) delivered by peer specialists. Each session will last up to 30 minutes.
  Interventions: Behavioral: Peer CBT Intervention
- Control (No Intervention): Women allocated to the observation-only control group will not receive any intervention.

INTERVENTIONS:
Behavioral: Peer CBT Intervention — Peer specialist delivery of cognitive behavioral therapy intervention over the phone.
  Arms: Peer CBT Intervention

SUMMARY:
Unintended pregnancy (UP), defined as a mistimed or unwanted pregnancy, is a significant and prevalent public health problem, particularly among low-income women. Over half of all pregnancies are reportedly unintended and UP has been linked to adverse health outcomes in mothers and their children. Correct and consistent use of effective contraception is the primary method to prevent UP. Research has shown that low self-esteem and elevated depressive symptoms increase women's risk for ineffective contraception use and, by extension, for UP. This project examines the feasibility and possible efficacy of reducing ineffective contraception using an intervention that addresses depressive symptoms and self concept among young, low-income, predominantly minority women at risk for UP. Traditional cognitive behavioral therapy (CBT) is effective in reducing depressive symptoms and improving self concept; but limited utilization, poor response, and low adherence to CBT is common among low-income and minority women. A more acceptable method for delivering CBT is needed for the target population. This project will use peer-specialists to deliver a CBT-based intervention to women at risk for UP. Because peer specialists are drawn from the same community as the target population and share some similar life experiences, the intervention may be more acceptable and effective than one offered by trained professionals.

This project will examine the effectiveness of a 9 week (8-session) peer-specialist led CBT-based intervention compared to an observational control condition to reduce depressive symptoms, improve self-esteem, and improve consistent contraceptive use to prevent UP. The weekly intervention sessions are delivered by telephone by a trained peer specialist. The study will evaluate the effectiveness of the intervention to improve consistent contraceptive use (primary outcome) and decrease depressive symptoms and increase self-esteem (secondary outcomes).

DETAILED DESCRIPTION:
This is a randomized controlled trial with one intervention group (peer-specialist led telephone-based CBT) and an observation only control group. There will be 3 measurement periods: baseline (pre-intervention), 10-week follow-up (post-intervention) and 14-week follow up. The 14-week follow up assesses the primary outcome (consistency of contraception use) and secondary outcomes (psychological symptoms and self-esteem), whereas the 10-week follow up assesses mediating variables (sexual self-efficacy, contraceptive self-efficacy, social support and coping). There is also a 4-week, mid-intervention assessment of outcomes designed to assess if there is a worsening of symptoms that needs to be addressed (e.g. referral for spike in depression or emergence of suicidal intent). This midterm evaluation also allows us to monitor the well-being of the control group, which has significantly less contact with project staff than the intervention group.

We will recruit 132 sexually active women from health care clinics (e.g., family planning, OB/GYN), with the aim of retaining at least 92 (46 per condition). Interested women will be consented and screened for eligibility in a private area of the clinics. They will be contacted by phone after consent to complete a structured, baseline questionnaire. After the baseline questionnaire, women will be randomly allocated to study conditions. Women will be randomized based on the randomization schedule established by the project biostatistician. Women allocated to the CBT intervention group will be mailed an intervention workbook and have their first telephone-based intervention session scheduled. The CBT intervention group will receive 8 telephone-based CBT intervention sessions (over 9 weeks) delivered by peer specialists. Each session will last up to 30 minutes. The control group will be an observation only control group (CTL group). They will not receive any intervention. The post-intervention and 1-month follow up questionnaires will also be collected via structured telephone interviews. Research staff who are collecting data will be blinded to study condition.

In addition to monitoring for worsening of psychological symptoms, procedures are in place for referring participants with worrisome increases in depression (i.e., >14 on the PHQ9) or suicidal intent to relevant mental health resources, including hospital emergency rooms and suicide hotlines for persons expressing suicidal intent. Further, the DSMB will be alerted so that they can monitor whether one condition appears to have an unusually high increase in symptoms, which might warrant stopping the trial for safety reasons. In addition, the researchers collecting data and the peer-specialists implementing the intervention will be engaged in weekly supervision with a clinical psychologist and have access to the study PI at all times. The project biostatistician will conduct all intention-to-treat (ITT) analyses using appropriate modern statistical approaches.

ELIGIBILITY:
Inclusion Criteria:

* female, aged 18-45, sexually active with a man in past 3 months, report inconsistent or no contraception use in the past 3 months, English speaking, own a smartphone, report subclinical to mild depressive symptoms in past two weeks (score 5 to 14 on PHQ-9)

Exclusion Criteria:

* pregnant, using Long Acting Reversible Contraceptives, sterilized, planning to get pregnant in the next 6 months, report acute suicide risk (assessed via the PHQ Follow-up Suicide Risk Assessment form or self-repot a suicide attempt in the past 6 months)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Consistent contraception use at 14-week follow-up | 14-week follow-up
  Categorical (yes/no). Self report of using birth control consistently in prior month with a male sexual partner.

SECONDARY OUTCOMES:
Change in mean level of depressive symptoms from baseline to 14-week follow-up | at 14-week follow-up
  9-item PHQ-9 Depressive Symptoms Scale. Self-report measure of depressive symptoms over the past two weeks. Each item is scored 0 (not at all) to 3 (nearly every day). Higher scores indicated greater depressive symptoms. The maximum score is 27. Symptom scores can be categorized by levels: 5-9 = minimal; 10-14 = mild; 15-19 moderately severed; 20+ = severe.
Change in mean level of self esteem from baseline to 14-week follow-up | at 14-week follow-up
  20-item State Self Esteem Scale. Self-report measure of state (current) self esteem, includes 3 subscales (performance, appearance, and social). Each item is scored 1 (not at all) to 5 (extremely). Items are coded such that higher scores indicated higher self esteem. A mean scale score is calculated, ranging from 1 to 5.

OTHER OUTCOMES:
Change in mean level of anxiety symptoms from baseline to 14-week follow-up | 14-week follow-up
  Exploratory secondary outcome measured with the 7-item Generalized Anxiety Disorder (GAD-7) scale. Each item is scored from 0 (not at all) to 3 (nearly every day). Items are summed with possible scores ranging from 0 to 21. Higher scores indicate more severe anxiety symptoms.
Change in mean level of somatic symptoms from baseline to 14-week follow-up | 14-week follow-up
  Exploratory secondary outcome measured with the 15-item Patient Health Questionnaire Somatic Symptom Scale (PHQ-15). Each item is scored from 0 (not bothered) to 2 (bothered a lot). Items are summed with possible scores ranging from 0 to 30. Higher scores indicate more severe somatic symptoms.
Change in mean level of perceived social support (belonging) from baseline to 10-week follow-up | 10-week follow-up
  Secondary outcome (mediator) measured with the 5-item General Mattering Scale. Items are scored from 0 (Not at all) to 4 (Very much). Items are summed with scores ranging from 0 to 20. Higher scores indicate a greater sense of mattering to others (belonging).
Change in mean level of sexual self-efficacy from baseline to 10-week follow-up | 10-week follow-up
  Secondary outcome (mediator) measured with 8 items representing the "Say No" subscale of Rosenthal's Sexual Self-Efficacy Scale. Each item is scored from 1 (Not at all sure) to 4 (Very sure). The mean level of self-efficacy is calculated with a range of 1 to 4.
Change in mean level of contraceptive self-efficacy from baseline to 10-week follow-up | 10-week follow-up
  Secondary outcome (mediator) measuring contraceptive self-efficacy. 5 items adapted from Lauby's self-efficacy measure for condom use. Items are scored from 1 (Not at all sure) to 4 (Very sure). Scores range from 5 to 20 and a higher score indicates greater perceived self-efficacy.
Change in mean level of coping from baseline to 10-week follow-up | 10-week follow-up
  Secondary outcome (mediator) measured with two subscales (8 items) of the COPE measure: planning (4 items) and positive reinterpretation and growth (4 items). Items are scored from 1 (Not at all) to 5 (Very much). Items for each subscale are summed with a possible score ranging from 4 to 20 for each subscale. Higher scores indicate more active coping efforts.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lepore, PHD, Principal Investigator — Temple University
Locations (1):
- Temple University School of Medicine OB/GYN, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There are no institutional resources (i.e., administrative and technical support) available at the end of the trial to support data sharing (e.g., review and respond to requests, store data and associated protocols, and deliver data and respond to queries about the data).